CLINICAL TRIAL: NCT01139593
Title: A Prospective Randomized Trial Comparing Qam With Qpm Daily Dosing in Assisted Reproductive Technologies
Brief Title: A Trial Comparing Qam With Qpm Dosing in Assisted Reproductive Technologies (ART)
Status: Completed | Type: Observational
Sponsor: Virginia Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Fady I. Sharara, M.D, Medical Director, Virginia Center for Reproductive Medicine
Other Study IDs: VCRM 5
Record Dates: First submitted 2010-06-06; First posted 2010-06-08 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: IVF; ICSI; gonadotropin; am dose; pm dose; pregnancy; implantation; live birth
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- morning dose: women undergoing IVF/ICSi taking their gonadotropin dose in the am
- evening dose: Women undergoing IVF/ICSI taking their gonadotropin in the evening

SUMMARY:
This is a prospective randomized trial comparing the outcome in women undergoing IVF/ICSI when taking their gonadotropin dosage in the morning (am) or evening (pm).

ELIGIBILITY:
Inclusion Criteria:

* women between 21-42 undergoing IVF

Exclusion Criteria:

* women > 45,
* women with one ovary,
* donor egg,
* surrogacy,
* FET cycles,
* uterine problems,
* large fibroids

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women between 21 and 44 years old
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Center for Reproductive Medicine, Reston, Virginia, United States